CLINICAL TRIAL: NCT05285046
Title: Phenotypic Profile and Molecular Mechanism of Resistance in Carbapenemase-producing Enterobacterales and Pseudomonas Aeruginosa Isolates From Brazilian Hospitals: Implications for the Introduction of IMIPENEM-RELEBACTAM
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: D'Or Institute for Research and Education (Other)
Responsible Party: Sponsor
Other Study IDs: 15054519.3.0000.5249B
Record Dates: First submitted 2022-02-28; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Bacterial Infections; Antibiotic Resistant Infection
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The global dissemination of carbapenem-resistant Enterobacteriaceae (CRE) and Pseudomonas aeruginosa (CRPA) are a significant threat to health care, especially for severely ill patients. Antibiotics currently used to treat CRE and CRPA infections are usually toxic and not very effective. Novel treatments include beta-lactamase inhibitors with broad-spectrum activity, among them IMI-REL. IMI-REL is a promising molecule due to the ability of REL to diminish carbapenem MICs to the susceptible range, potentially restoring the activity of this potent drug. However, few studies have systematically examined IMI-REL activity against a diverse clinical collection of CRE and CRPA strains, in particular from a region where the resistance is high, and the main mechanisms are in general unknown (Brazil- Latin America). As the use of molecular diagnostics becomes increasingly available in clinical settings, it is crucial to identify molecular markers predicting antimicrobial efficacy to guide therapeutic decision-making. In the present study, we will acess different species of CRE and CRPA from clinically relevant isolates to determine if the species, clonal lineage, and resistance gene profile, have influence to the response to IMI-REL.

DETAILED DESCRIPTION:
Prospective evaluation of 150 (one hundred and fifty) Enterobacterales and 100 (one hundred) Pseudomonas aeruginosa isolates from 12 hospitals in the city of Rio de Janeiro. A sequential number of isolates per unit will be selected considering the inclusion criteria of resistance to carbapenem, only one isolate per patient will be evaluated. The isolate will be identified in genus and species by the VITEK® MS MALDI-TOF (bioMérieux - France) mass spectrometry methodology from bloodstream isolates and respiratory specimens.

The detection of carbapenemase production by rapid colorimetric method will be performed using the RAPIDEC® Carba NP test (bioMérieux - France). The isolates that present positive carbapenemase test by colorimetric method will be submitted to the PCR extended-spectrum beta-lactamase and carbapenemase gene characterization test for the following genes: blaSHV, blaCTX-M, KPC, NDM, VIM, IMP, SME , NMC / IMI, GES, GIM, SMP, IMP, OXA 23, OXA 24, OXA 48, OXA 51 and OXA 58.

After characterization of the carbapenemase-producing genes, isolates possessing the Class A and D carbapenemase gene, it will be evaluated the susceptibility profile of imipenem-relebactam using BMD (Broth Microdilution) to determine the minimum inhibitory concentration and its respective sensitivity and resistance criteria using recent CLSI MIC breakpoints - M100, 29th Ed (Clinical and Laboratory Standards Institute - 2020) and EUCAST Version 10.0 (European Committee on Antimicrobial Susceptibility Testing V 10.0). Isolates showing positive results for carbapenemase production, but with negative PCR results for the genes described above, will be further investigated for the likely presence of other carbapenemase producing genes or other mechanisms of resistance to carbapenem antibiotics. For the study and evaluation of the genetic diversity of the isolates, the Multilocus Sequence Typing (MLST) methodology will be used. Isolates that show simultaneous resistance to carbapenems, polymyxin B and fluoroquinolones will be subjected to next generation sequencing (NGS) for further evaluation of other genes or mechanisms associated with antibiotic resistance or virulence markers.

ELIGIBILITY:
Inclusion Criteria:

* Microbiologics analysis indicating carbapenem resistance

Exclusion Criteria:

* Microbiologics analysis indicating Negative class A and D cabapenemase gene

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will evaluate prospectively 150 (one hundred and fifty) Enterobacterales and 100 (one hundred) Pseudomonas aeruginosa isolates from 12 hospitals in Rio de Janeiro.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-10-30 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Susceptibility profile of imipenem-relebactam | immediately after the analysis.
  Evaluation of the susceptibility profile of imipenem-relebactam in isolates possessing the Class A and D carbapenemase gene.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Bozza, PhD, Principal Investigator — D'Or Institute for Research and Education (IDOR)
Locations (1):
- D'Or Institute for Research and Education (IDOR), Rio de Janeiro, Brazil